CLINICAL TRIAL: NCT00442702
Title: An Open-label, Randomized, Multi-center, Parallel Group Non-inferiority Study of Subcutaneous Injections of RO0503821 Given Once Monthly vs. Darbepoetin Alfa Given According to Local Label in Patients With Chronic Kidney Disease Who Are Not on Dialysis.
Brief Title: A Study of Subcutaneous Mircera in Patients With Chronic Kidney Disease, Not on Dialysis.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BH20051
Record Dates: First submitted 2007-03-01; First posted 2007-03-02 (Estimated); Results first posted 2011-10-03 (Estimated); Last update posted 2011-12-19 (Estimated); Status verified 2011-12

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — continuous erythropoietin receptor activator; Darbepoetin alfa

ARMS (2):
- Mircera (Experimental): Participants received Mircera by subcutaneous injection once every month during the dose titration (7 months) and evaluation period (2 months). The starting dose was based on the weekly dose of darbepoetin alfa administered prior to the switch to Mircera, and was either 120, 200 or 360 µg Mircera per month. The dose was then adjusted to maintain Hemoglobin levels within the defined target range and also according to the need for red blood cell transfusions (due to worsening anemia), or for toxicity related to Mircera.
  Interventions: Drug: Mircera
- Darbepoetin alfa (Active Comparator): Participants continued to receive the same dose of darbepoetin alfa as before screening by subcutaneous injection once every week, once every 2 weeks or once every month as per local labeling during the dose titration (7 months) and the evaluation period (2 months).
  Interventions: Drug: Darbepoetin alfa

INTERVENTIONS:
Drug: Mircera — Starting dose of 120, 200 and 360 micrograms administered by subcutaneous injection once a month.
  Other Names: RO0503821; Methoxy polyethylene glycol-epoetin beta
  Arms: Mircera
Drug: Darbepoetin alfa — As prescribed, subcutaneous injection once every week, once every 2 weeks or once every month as per local labeling specifications.
  Other Names: Aranesp®
  Arms: Darbepoetin alfa

SUMMARY:
This 2 arm study will compare the efficacy and safety of Mircera and darbepoetin alfa in the treatment of anemia in patients with chronic kidney disease who are not on dialysis and who are receiving subcutaneous darbepoetin alfa maintenance therapy. Patients will be randomized either to remain on darbepoetin alfa therapy as per local label, or to switch to monthly subcutaneous Mircera, at a starting dose of 120, 200 or 360 micrograms, depending on the weekly dose of darbepoetin alfa administered prior to the first dose of Mircera. The anticipated time on study treatment is 3-12 months, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* chronic kidney disease, not requiring dialysis;
* receiving darbepoetin alfa maintenance therapy for >=8 weeks before screening, and during screening/baseline period.

Exclusion Criteria:

* overt gastrointestinal bleeding within 8 weeks before screening, or during screening/baseline period;
* transfusion of red blood cells within 8 weeks before screening, or during screening/baseline period;
* active malignant disease;
* previous treatment with Mircera.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2007-09; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (86):
- United States (11):
  - Granada Hills, California
  - Lauderdale Lakes, Florida
  - Augusta, Georgia
  - Mineola, New York
  - Orchard Park, New York
  - Raleigh, North Carolina
  - Oregon City, Oregon
  - Providence, Rhode Island
  - Chattanooga, Tennessee
  - Salem, Virginia
  - Morgantown, West Virginia
- Australia (5):
  - Adelaide
  - Gosford
  - Lismore
  - Reservoir
  - Richmond
- Belgium (2):
  - Aalst
  - Roeselare
- Canada (6):
  - Calgary, Alberta
  - St. John's, Newfoundland and Labrador
  - Kingston, Ontario
  - Mississauga, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
- Czechia (2):
  - Mariánské Lázně
  - Prague
- France (7):
  - La Tronche
  - Nantes
  - Orléans
  - Paris
  - Rennes
  - Saint-Priest-en-Jarez
  - Strasbourg
- Germany (8):
  - Bad Hersfeld
  - Bad König
  - Berlin
  - Bonn
  - Coburg
  - Demmin
  - Dortmund
  - München
- Hungary (8):
  - Baja
  - Budapest
  - Esztergom
  - Hódmezővásárhely
  - Kalocsa
  - Kecskemét
  - Szigetvár
  - Vác
- Israel (5):
  - Hadera
  - Jerusalem
  - Kfar Saba
  - Nahariya
  - Rehovot
- Italy (12):
  - Brescia
  - Chieti
  - Ferrara
  - Genova
  - La Spezia
  - Lecco
  - Lodi
  - Palermo
  - Pavia
  - Prato
  - Roma
  - S Fermo Della Battaglia
- Poland (8):
  - Gdansk
  - Katowice
  - Lodz
  - Radom
  - Rzeszów
  - Sieradz
  - Szczecin
  - Warsaw
- Spain (8):
  - A Coruña
  - Barcelona
  - Ciudad Real
  - L'Hospitalet de Llobregat
  - Lleida
  - Madrid
  - Málaga
  - Partida La Ceñuela. Torreviej
- United Kingdom (4):
  - Belfast
  - Birmingham
  - Bradford
  - Exeter

REFERENCES:
- [Derived] Chung EY, Palmer SC, Saglimbene VM, Craig JC, Tonelli M, Strippoli GF. Erythropoiesis-stimulating agents for anaemia in adults with chronic kidney disease: a network meta-analysis. Cochrane Database Syst Rev. 2023 Feb 13;2(2):CD010590. doi: 10.1002/14651858.CD010590.pub3. PMID 36791280

RESULTS

PARTICIPANT FLOW:
Groups:
- Darbepoetin Alfa: Participants continued to receive the same dose of darbepoetin alfa by subcutaneous injection once every week, once every 2 weeks or once every month as per local labeling during the dose titration (7 months) and the evaluation period (2 months).
Period: Titration Period
Arm/Group | Mircera | Darbepoetin Alfa
Started | 114 | 114
Safety Population | 115 (One patient was randomized to darbepoetin alfa but treated by mistake with Mircera) | 113
Completed | 102 | 111
Not Completed | 12 | 3
Not completed — Adverse Event | 2 | 0
Not completed — Death | 3 | 2
Not completed — Insufficient Therapeutic Response | 1 | 0
Not completed — Refused Treatment | 4 | 1
Not completed — Failure to return | 1 | 0
Not completed — Hospitalized in another hospital | 1 | 0
Period: Evaluation Period
Arm/Group | Mircera | Darbepoetin Alfa
Started | 102 | 111
Completed | 97 | 107
Not Completed | 5 | 4
Not completed — Adverse Event | 1 | 0
Not completed — Death | 1 | 1
Not completed — Insufficient Therapeutic Response | 1 | 0
Not completed — Refused treatment | 1 | 1
Not completed — Renal transplant | 0 | 1
Not completed — Failure to return | 1 | 0
Not completed — Site closure | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mircera | Darbepoetin Alfa | Total
Number analyzed (Participants) | 114 | 114 | 228
Age Continuous [Mean (Standard Deviation); unit: years] | 71.3 (11.03) | 69.6 (14.02) | 70.4 (12.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 66 | 132
  Male | 48 | 48 | 96

OUTCOME MEASURES:

1. Primary Outcome: Change in Hemoglobin (Hb) Concentration From Baseline to the Evaluation Period
Description: A time adjusted average baseline hemoglobin (Hb) concentration was calculated using the trapezoid rule from all available Hb measurements taken during the baseline period. The average evaluation period Hb concentration for each individual was calculated using the same method, from all their available measurements taken during the two month evaluation period. The change in Hb concentration between the baseline and evaluation periods was calculated by subtracting the baseline Hb from the evaluation period Hb. All blood samples for Hb measurements were taken prior to study drug administration.
Time Frame: Baseline (measurements at Week -4, Week -2 and Day 1) and Evaluation Period (Months 8 and 9; measurements twice a month and at the final visit).
Population: Per Protocol population consisted of all randomized patients who had received at least one dose of trial medication and who have no major protocol violation. Data missing at the end of the evaluation period were handled using the last observation carried forward method (LOCF).
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Mircera | Darbepoetin Alfa
Number analyzed (Participants) | 91 | 99
g/dL
  Baseline Hb | 11.29 (0.382) | 11.33 (0.397)
  Change from baseline | 0.15 (0.899) | -0.03 (0.693)

2. Secondary Outcome: Change in Hemoglobin Concentration From Baseline Over Time
Time Frame: From Baseline to 9 months; blood samples for hemoglobin measurements were taken twice a month, at each study visit.
Population: Intent-to-treat population, including all randomized patients. "n" refers to the number of patients for whom data was available at each time point.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Mircera | Darbepoetin Alfa
Number analyzed (Participants) | 114 | 114
g/dL
  Baseline [n=114, 114] | 11.27 (0.390) | 11.31 (0.393)
  Change at 0.5 Months [n=113, 114] | 0.29 (0.737) | 0.03 (0.490)
  Change at 1 Month [n=114, 113] | 0.34 (0.813) | 0.06 (0.575)
  Change at 1.5 Months [n=111, 113] | 0.45 (0.866) | 0.11 (0.599)
  Change at 2 Months [n=112, 112] | 0.27 (0.897) | 0.02 (0.716)
  Change at 2.5 Months [n=110, 112] | 0.45 (0.924) | 0.16 (0.673)
  Change at 3 Months [n=111, 112] | 0.23 (1.010) | 0.10 (0.602)
  Change at 3.5 Months [n=108, 108] | 0.18 (1.095) | 0.05 (0.675)
  Change at 4 Months [n=109, 110] | 0.05 (0.893) | 0.00 (0.681)
  Change at 4.5 Months [n=104, 108] | 0.18 (0.940) | 0.13 (0.699)
  Change at 5 Months [n=108, 111] | -0.03 (0.897) | -0.07 (0.757)
  Change at 5.5 Months [n=105, 110] | 0.15 (0.922) | -0.03 (0.729)
  Change at 6 Months [n=103, 111] | -0.05 (0.988) | -0.06 (0.820)
  Change at 6.5 Months [n=100, 110] | 0.06 (1.087) | 0.04 (0.817)
  Change at 7 Months [n=102, 111] | 0.03 (1.008) | -0.00 (0.842)
  Change at 7.5 Months [n=99, 110] | 0.12 (1.166) | -0.00 (0.873)
  Change at 8 Months [n=100, 108] | -0.04 (1.198) | -0.12 (0.905)
  Change at 8.5 Months [n=97, 107] | 0.14 (1.256) | 0.02 (0.766)
  Change at 9 Months [n=94, 101] | 0.07 (1.045) | -0.06 (0.956)

3. Secondary Outcome: Number of Participants With Red Blood Cell (RBC) Transfusions
Description: Red blood cell (RBC) transfusions could be given during the treatment period in case of medical need, i.e., in severely anemic patients with recognized symptoms or signs of anemia (e.g., in patients with acute blood loss, with severe angina, or whose Hemoglobin decreased to critical levels). The number of participants who had at least one red blood cell transfusion during the entire study, during the Titration Period and during the Evaluation Period is presented. Participants who received more than one transfusion within a defined period are only counted once.
Time Frame: From randomization to Month 9
Population: Safety population included all randomized patients who received at least one dose of trial medication and a safety follow-up, according to the treatment received.
Measure: Number; unit: participants
Arm/Group | Mircera | Darbepoetin Alfa
Number analyzed (Participants) | 115 | 113
participants
  Entire Study | 9 | 3
  Titration Period | 5 | 1
  Evaluation Period | 5 | 2

4. Secondary Outcome: Participants With Adverse Events
Description: Adverse events were collected during the treatment period (from the first treatment dose) up to 30 days after last dose or at least until the date of last contact if the date of last contact occurred after the specified 30 day period.
Time Frame: Randomization to Month 10 (final visit)
Population: Safety population
Measure: Number; unit: participants
Arm/Group | Mircera | Darbepoetin Alfa
Number analyzed (Participants) | 115 | 113
participants
  Any adverse event | 102 | 88
  Fatal Adverse event | 4 | 3
  Serious adverse event | 41 | 23
  Adverse event leading to withdrawal | 3 | 0

ADVERSE EVENTS:
Time Frame: All adverse events that occurred from the first treatment dose were summarized. Adverse events were included up to 30 days after last dose or at least until the date of last contact if the date of last contact occurred after the specified 30 day period.
Description: Safety population was used for analysis.
Arm/Group | Mircera | Darbepoetin Alfa
Serious Adverse Events (participants affected / at risk) | 41/115 | 23/113
Other Adverse Events (participants affected / at risk) | 59/115 | 49/113
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mircera (N=115) | Darbepoetin Alfa (N=113)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 2 | 1
ATRIAL FIBRILLATION (Cardiac disorders) | 1 | 1
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1 | 0
AORTIC VALVE DISEASE MIXED (Cardiac disorders) | 1 | 0
ARRHYTHMIA (Cardiac disorders) | 1 | 0
ATRIAL FLUTTER (Cardiac disorders) | 1 | 0
BRADYCARDIA (Cardiac disorders) | 0 | 1
CARDIAC FAILURE (Cardiac disorders) | 0 | 1
CARDIOGENIC SHOCK (Cardiac disorders) | 1 | 0
CORONARY ARTERY DISEASE (Cardiac disorders) | 1 | 0
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 | 0
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 1 | 0
SICK SINUS SYNDROME (Cardiac disorders) | 1 | 0
SILENT MYOCARDIAL INFARCTION (Cardiac disorders) | 1 | 0
PNEUMONIA (Infections and infestations) | 2 | 1
RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 | 0
BRONCHOPNEUMONIA (Infections and infestations) | 1 | 0
CORYNEBACTERIUM SEPSIS (Infections and infestations) | 0 | 1
GASTROENTERITIS (Infections and infestations) | 1 | 0
INFECTED SKIN ULCER (Infections and infestations) | 1 | 0
NEUROLOGICAL INFECTION (Infections and infestations) | 1 | 0
OSTEOMYELITIS (Infections and infestations) | 1 | 0
POST PROCEDURAL INFECTION (Infections and infestations) | 1 | 0
URINARY TRACT INFECTION (Infections and infestations) | 0 | 1
FLUID OVERLOAD (Metabolism and nutrition disorders) | 1 | 1
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 | 2
DEHYDRATION (Metabolism and nutrition disorders) | 1 | 0
DIABETES MELLITUS INADEQUATE CONTROL (Metabolism and nutrition disorders) | 0 | 1
FLUID RETENTION (Metabolism and nutrition disorders) | 1 | 0
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 1 | 0
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 | 0
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 | 1
ATAXIA (Nervous system disorders) | 1 | 0
HEADACHE (Nervous system disorders) | 1 | 0
NERVE ROOT COMPRESSION (Nervous system disorders) | 0 | 1
PARTIAL SEIZURES (Nervous system disorders) | 1 | 0
SCIATICA (Nervous system disorders) | 1 | 0
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 | 1
VERTEBROBASILAR INSUFFICIENCY (Nervous system disorders) | 0 | 1
RENAL IMPAIRMENT (Renal and urinary disorders) | 5 | 0
RENAL FAILURE CHRONIC (Renal and urinary disorders) | 2 | 1
CALCULUS URETERIC (Renal and urinary disorders) | 0 | 1
PANCREATITIS ACUTE (Gastrointestinal disorders) | 2 | 0
COLITIS ISCHAEMIC (Gastrointestinal disorders) | 1 | 0
DIARRHOEA (Gastrointestinal disorders) | 1 | 0
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
HIATUS HERNIA (Gastrointestinal disorders) | 1 | 0
RECTAL POLYP (Gastrointestinal disorders) | 1 | 0
LOWER LIMB FRACTURE (Injury, poisoning and procedural complications) | 2 | 0
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
PELVIC FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
VERTIGO (Ear and labyrinth disorders) | 1 | 2
ANGIOSARCOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
COLON CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
ARTERIOSCLEROSIS (Vascular disorders) | 0 | 1
EXTREMITY NECROSIS (Vascular disorders) | 1 | 0
HYPERTENSION (Vascular disorders) | 0 | 1
NON-CARDIAC CHEST PAIN (General disorders) | 0 | 1
OEDEMA PERIPHERAL (General disorders) | 1 | 0
CHOLECYSTITIS (Hepatobiliary disorders) | 1 | 0
CHOLELITHIASIS (Hepatobiliary disorders) | 1 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 | 0
PATHOLOGICAL FRACTURE (Musculoskeletal and connective tissue disorders) | 1 | 0
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 | 1
SKIN ULCER (Skin and subcutaneous tissue disorders) | 2 | 0
NEPHROGENIC ANAEMIA (Blood and lymphatic system disorders) | 1 | 0
CATARACT (Eye disorders) | 0 | 1
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Mircera (N=115) | Darbepoetin Alfa (N=113)
HYPERTENSION (Vascular disorders) | 30 | 20
NASOPHARYNGITIS (Infections and infestations) | 7 | 13
URINARY TRACT INFECTION (Infections and infestations) | 10 | 4
RENAL IMPAIRMENT (Renal and urinary disorders) | 13 | 12
DIARRHOEA (Gastrointestinal disorders) | 5 | 8
CONSTIPATION (Gastrointestinal disorders) | 6 | 3
OEDEMA DUE TO RENAL DISEASE (General disorders) | 6 | 7
HYPERPARATHYROIDISM SECONDARY (Endocrine disorders) | 8 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 6 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.